CLINICAL TRIAL: NCT01580995
Title: HSV-1 Suppression in HCV Infected Veterans Who Are Seronegative for HSV-2
Brief Title: Herpes Simplex Type 1 Suppression in Hepatitis C
Acronym: HSV1/HCV
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CLIN-001C-10F
Record Dates: First submitted 2012-04-13; First posted 2012-04-19 (Estimated); Results first posted 2016-09-21 (Estimated); Last update posted 2016-09-21 (Estimated); Status verified 2016-08

CONDITIONS: Chronic Hepatitis C Infection
Keywords: Chronic hepatitis C infection
MeSH Terms: interventions — Valacyclovir

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Valacyclovir (Experimental): Valacyclovir 500 mg po bid
  Interventions: Drug: Valacyclovir
- Placebo (Placebo Comparator): Matching placebo twice daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Valacyclovir — Valacyclovir 500 mg po bid
  Arms: Valacyclovir
Drug: Placebo — Placebo tablet twice daily
  Arms: Placebo

SUMMARY:
The purpose of this study is to examine the effects of valacyclovir in patients who have chronic hepatitis C, antibodies to herpes simplex type 1 infection but do not have antibodies to herpes simplex type 2 infection. Herpes simplex type 1 infection commonly causes cold sores or fever blisters, also known as herpes labialis, but most persons do not have any symptoms at all. Valacyclovir is a medication which is approved by the Food and Drug administration to treat herpes labialis. Valacyclovir has not been approved to treat chronic hepatitis C infection.

The study will take 16 weeks. Participants will be assigned to take either the study drug, valacyclovir, or a sugar pill that looks exactly like valacyclovir. The researchers and patients will not know which medication they are receiving. Study visits will occur every two weeks and will take approximately 30-45 minutes. All study visits will occur at the G.V. Sonny Montgomery VA Medical Center in Jackson, Mississippi.

DETAILED DESCRIPTION:
This is a randomized double-blind placebo-controlled clinical trial evaluating the effect of 500 mg valacyclovir twice daily on HCV viral load in HSV-1/HCV co-infected patients seronegative for HSV-2. Potential participants will be recruited from the Jackson VAMC viral hepatitis clinics. Eligible individuals will be invited to enroll in the study in a noncoercive manner. Study personnel will obtain full informed consent.

Using a computer generation randomization scheme, patients will be randomized 1:1 in blocks of 4 to receive valacyclovir 500 mg po twice daily or matching placebo. Patients will be counseled on the signs and symptoms of herpes labialis and genital herpes and complete a questionnaire to document medical/social history. Venipuncture will be performed every four weeks (i.e., at every other follow-up visit) to monitor complete blood cell count, liver function tests, serum levels of hepatitis C RNA and Herpeselect IgG HSV-2 ELISA. A de-identified baseline serum sample will be collected and stored in VA approved research space for future testing. At each visit, pill-count and tolerability of medications will be assessed. Patients will be asked about signs or symptoms of genital herpes. Data will be kept in a study chart labeled with the participant's coded study number in a locked office. Information from each study visit will be recorded into the chart by the PI or RA and entered into an encrypted database on a secure VA server. Baseline characteristics of the placebo and intervention group will be compared using appropriate parametric tests. HCV viral loads will be log10 transformed and analyzed using an intention to treat model.

ELIGIBILITY:
Inclusion Criteria:

* Chronic hepatitis C infection with a detectable HCV RNA in the serum on two occasions, 6 months apart
* Focus HSV-2 IgG negative and Focus HSV-1 IgG positive, using manufacturer's cut-offs

Exclusion Criteria:

* Antiherpes or immunomodulatory therapy during the past 30 days,
* HIV or chronic hepatitis B infection,
* Decompensated liver disease (ascites, hepatic encephalopathy, coagulopathy, jaundice/icterus),
* Creatinine clearance <50 ml/min.,
* Female subject who is pregnant or nursing,
* Gastrointestinal disorder which might result in malabsorption of valacyclovir,
* History of erythema multiforme major, thrombotic thrombocytopenia purpura or hemolytic uremic syndrome,
* Allergy to valacyclovir or related drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2012-04; Primary Completion 2014-12 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary J Burton, MD, Principal Investigator — G.V. (Sonny) Montgomery VA Medical Center, Jackson, MS
Locations (1):
- G.V. (Sonny) Montgomery VA Medical Center, Jackson, MS, Jackson, Mississippi, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Valacyclovir | Placebo
Started | 10 | 9
Completed | 8 | 7
Not Completed | 2 | 2
Not completed — Lost to Follow-up | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Valacyclovir | Placebo | Total
Number analyzed (Participants) | 10 | 9 | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 9 | 19
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 55 (2) | 57 (3) | 56 (2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 10 | 9 | 19
Region of Enrollment [Number; unit: participants]
  United States | 10 | 9 | 19

OUTCOME MEASURES:

1. Primary Outcome: Change in HCV RNA Viral Load
Description: Measure change in HCV RNA viral load in treatment group as compared with placebo
Time Frame: Baseline, 12 weeks
Population: patients who completed 12 weeks of follow up
Measure: Mean (Standard Deviation); unit: log(IU/mL)
Arm/Group | Valacyclovir | Placebo
Number analyzed (Participants) | 8 | 7
log(IU/mL) | .24 (.20) | .08 (.01)
Statistical Analysis 1: Comparison: Valacyclovir vs Placebo; Test type: Superiority or Other; p = 0.05, Fisher Exact

ADVERSE EVENTS:
Arm/Group | Valacyclovir | Placebo
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/9
Other Adverse Events (participants affected / at risk) | 0/10 | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No